CLINICAL TRIAL: NCT02642627
Title: The Use of Bellafill for Atrophic Acne Scar Correction in the Full Facial Area
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suneva Medical, Inc. (Industry)
Collaborators: ethica Clinical Research Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SUN-1504
Record Dates: First submitted 2015-12-28; First posted 2015-12-30 (Estimated); Results first posted 2020-04-06 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2019-09

CONDITIONS: Atrophic Acne Scarring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bellafill Injections (Experimental): Correctable acne scars will be individually identified and only scars that the Investigator determines to be correctable will receive study treatment. All eligible scars within the treatment area will be treated. Bellafill will be injected using a standard tunneling technique whereby the filler is injected in a retrograde manner utilizing several passes until the scar reaches a desired level of correction. A touch-up treatment is allowed if additional treatment is required to achieve optimal correction.
  Interventions: Device: Bellafill

INTERVENTIONS:
Device: Bellafill

SUMMARY:
This is an open-label, multicenter, prospective pilot study assessing the efficacy and safety of Bellafill for correction of distensible atrophic acne scars in the full facial area. All enrolled subjects will receive initial treatment with Bellafill, as well as touch-up treatments (if necessary to achieve optimal correction). Subjects will be evaluated at Screening (Month -1), Day 0 (Baseline) Month 1, Month 4, and Month 7.

DETAILED DESCRIPTION:
Correctable acne scars will be individually identified and only scars that the Investigator determines to be correctable will receive study treatment. All eligible scars within the treatment area will be treated.

Bellafill should be injected using a standard tunneling technique whereby the filler is injected in a retrograde manner utilizing several passes until the scar reaches a desired

level of correction. A touch-up treatment is allowed if additional treatment is required to achieve optimal correction.

Treatment Area

There will be four "quadrants" of the face where treatment is allowed and grading will occur. The glabellar, nose and upper lip areas are not to be treated:

* The glabellar "no treatment" zone is defined as the area between the mid-pupillary lines up to 2 cm above the highest point of the eyebrow. This area will not receive treatment;
* The no treatment area of the nose extends from the nasal bridge (and is contiguous with the glabellar no treatment zone) to the nasal sill and laterally to the cheek;
* The upper lip will be defined as the area from the vermillion border of the upper lip to the nasal sill superiorly and the nasolabial fold laterally;
* The face is split at the midline of the forehead and the chin and where the nose meets the cheek, creating two halves. Each half is then divided into upper and lower quadrants by a line extending from the lateral canthus to the superior junction of the pinna and the cheek.

Each quadrant will be graded individually and receive a separate grade. The no treatment zones of the glabella, nose and upper lip should be respected as they have been selected to maximize the safety of the subject. A "touch-up treatment" is permitted at study Visit 3 (Month 1). The Investigator will evaluate each lesion and determine if a treated scar is undercorrected and whether additional improvement could be obtained with a touch-up treatment.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient, male or female subjects of any race, 21 years of age or older. Female subjects of childbearing potential must have a negative urine pregnancy test result at Baseline and practice a reliable method of contraception throughout the study.
* Negative response to the Bellafill Skin Test.
* Presence of ≥4 distensible atrophic acne scars (treatment scars) in in the facial area.
* Subject desires correction of his/her atrophic acne scarring.
* All Fitzpatrick skin types are eligible.
* Willing to withhold additional aesthetic therapies to the proposed treatment area (e.g., other soft tissue fillers such as hyaluronic acid, and/or any resurfacing procedures (as described in Protocol Section 5.4) for the duration of the study.
* Able to follow study instructions and likely to complete all required visits, as assessed by the Investigator.
* Sign an IRB-approved Informed Consent Form, Photographic Release Form, and the Authorization for Use and release of Health and Research Study Information (HIPAA) Form prior to any study-related procedures being performed.

Exclusion Criteria:

* Female subjects that are pregnant (positive urine pregnancy test), breast-feeding, or who are of childbearing potential and not practicing a reliable method of birth control.
* Undergone facial treatments with any prohibited treatment/procedures and/or use of any other prohibited treatment/procedure within certain time periods as listed in Protocol Section 5.4.
* Excisional facial surgery (such as Blepharoplasty, Face Lift, Rhinoplasty) of the face less than 6 months prior to study enrollment or plans for facial surgery during the study.
* History of bleeding disorders.
* Presence of any skin pathology or condition that could interfere with the evaluation of the treatment areas, worsen due to the proposed treatment or require interfering topical, systemic or surgical therapy.
* Recent or current history of inflammatory skin disease, infection, cancerous/pre-cancerous lesion, unhealed wound or clinically significant acne in the proposed treatment areas. Clinically significant acne is defined as a patient whom has ≥3 active inflammatory acne lesions in the treatment areas.
* History of systemic granulomatous diseases active or inactive (e.g., Sarcoid, Wegeners, TB) or connective tissue diseases (e.g., lupus, dermatomyositis).
* Hypertrophic acne scars, any evidence of keloid scarring in the treatment area.
* Known hypersensitivity or previous allergic reaction to any of the components of the study device (including lidocaine or any amide-based anesthetic), or has a history of allergies to any bovine collagen products, including but not limited to injectable collagen, collagen implants, hemostatic sponges, and collagen-based sutures.
* Undergone or be planning to undergo desensitization injections to meat products.
* Unable to communicate or cooperate with the Investigator due to a language barrier (non-English speaking), poor mental development, or impaired cerebral function.
* Evidence of alcohol or drug abuse (Investigator opinion), or history of poor cooperation, non-compliance with medical treatment, or unreliability.
* Use of an investigational device, biologic or drug in the past 30 days, or be currently participating in an experimental drug, biologic or device trial.
* Exhibits additional physical attributes which prevent the assessment or treatment of the atrophic scars, as judged by the Investigator, such as excessive hair, traumatic or surgical scars, excessive hyperpigmentation in the treatment area, etc.
* Has a condition or be in a situation that, in the Investigator's opinion, may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study.
* An employee (or a relative of an employee) of the Investigator, Sponsor or representative of the Sponsor.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-11-18 (Actual); Primary Completion 2017-01-27 (Actual); Study Completion 2017-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Seretta, Study Director — Suneva Medical
Locations (1):
- Call Suneva for Info, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Joseph JH, Shamban A, Eaton L, Lehman A, Cohen S, Spencer J, Bruce S, Grimes P, Tedaldi R, Callender V, Werschler P. Polymethylmethacrylate Collagen Gel-Injectable Dermal Filler for Full Face Atrophic Acne Scar Correction. Dermatol Surg. 2019 Dec;45(12):1558-1566. doi: 10.1097/DSS.0000000000001863. PMID 30829754

RESULTS

PARTICIPANT FLOW:
Groups:
- Bellafill Injections: Correctable acne scars will be individually identified and only scars that the Investigator determines to be correctable will receive study treatment. All eligible scars within the treatment area will be treated. Bellafill will be injected using a standard tunneling technique whereby the filler is injected in a retrograde manner utilizing several passes until the scar reaches a desired level of correction. A touch-up treatment is allowed if additional treatment is required to achieve optimal correction.
  Bellafill
Period: Overall Study
Arm/Group | Bellafill Injections
Started | 42
Completed | 39
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Bellafill Injections
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.38 (12.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 26
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 42

OUTCOME MEASURES:

1. Primary Outcome: Change on the Acne Scar Assessment Scale (ASAS)
Description: A validated 5-point static scale assessing physician impression of acne scar severity. The total range on the scale is 1-5 (1= Clear and 5 = Severe) Clear: No depressions are seen in the treatment area. Macular discoloration may be seen.
  Very Mild: A single depression is easily noticeable with direct lighting (deep). Most or all of the depressions seen are only readily apparent with tangential lighting (shallow).
  Mild: A few to several, but less than half of all the depressions are easily noticeable with direct lighting (deep). Most of the depressions seen are only readily apparent with tangential lighting (shallow).
  Moderate: More than half of the depressions are apparent with direct lighting (deep).
  Severe: All or almost all the lesions can be seen with direct lighting (deep)
Time Frame: Month 1, 4 and 7
Population: The overall number of participants was all subjects enrolled in the clinical trial. The number analyzed includes the number of participants with available data for each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bellafill Injections
Number analyzed (Participants) | 42
units on a scale
  Month 1 | 3.33 (0.78)
  Month 4: number analyzed (Participants) | 39
  Month 4 | 2.19 (0.65)
  Month 7: number analyzed (Participants) | 39
  Month 7 | 2.20 (0.67)

2. Secondary Outcome: Adverse Events
Description: Throughout the course of the study, all AEs will be monitored and reported through the CRF. All AEs occurring after study device administration were followed until the event has resolved or stabilized or until follow-up was no longer possible.
Time Frame: month 7
Measure: Number; unit: adverse events
Arm/Group | Bellafill Injections
Number analyzed (Participants) | 42
adverse events
  All Adverse Events | 6
  Treatment Related Adverse Events | 2

ADVERSE EVENTS:
Time Frame: 7 months
Arm/Group | Bellafill Injections
All-Cause Mortality (participants affected / at risk) | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42
Other Adverse Events (participants affected / at risk) | 6/42
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bellafill Injections (N=42)
Bruising (Skin and subcutaneous tissue disorders) | 2 (2)
Injection Site hemorrhage (Skin Test) (Skin and subcutaneous tissue disorders) | 1 (1)
Injection Site Pain (General disorders) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1)
Contact Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2015-10-05): https://cdn.clinicaltrials.gov/large-docs/27/NCT02642627/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2015-08-28): https://cdn.clinicaltrials.gov/large-docs/27/NCT02642627/Prot_SAP_001.pdf